CLINICAL TRIAL: NCT04766580
Title: Placebo Effect in Children With Attention Deficit Disorder and/or Hyperactivity Disorder
Brief Title: Attention and Pain in Children With and Without Attention Deficit and/or Hyperactivity Disorder
Acronym: ADE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Guillaume Léonard, Principal Investigator, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-3357
Record Dates: First submitted 2021-02-17; First posted 2021-02-23 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Placebo Effect; Nocebo Effect; Pain
Keywords: Placebo; Nocebo; Attention; Pain; Children; Imaging
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Pain | interventions — Nocebo Effect

STUDY DESIGN:
Intervention Model Description: All the participants will take "two medications" (which are all placebos). The order of the "medications" are randomized.
Who Masked: Participant
Masking Description: The participants think they are taking two medications (if not in the "control group"), but the care provider and investigators know that only placebos (a placebo and a nocebo) are given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with ADHD group (Experimental): The same protocol is used for both groups
  Interventions: Behavioral: Placebo and nocebo effect
- Children with no ADHD group (Active Comparator): The same protocol is used for both groups
  Interventions: Behavioral: Placebo and nocebo effect

INTERVENTIONS:
Behavioral: Placebo and nocebo effect — The intervention focuses on the speech and instructions given with each placebo (positive for the placebo effect and negative for the nocebo effect)
  Other Names: Pygmalion effect

SUMMARY:
In Quebec, there has been an important increase of Attention Deficit Hyperactivity Disorder (ADHD) diagnosis since 2015. ADHD symptoms, related to behavioural and/or concentration difficulties, are very similar to other disorders symptoms, such as anxiety and depression, and have a significant impact on students' academic success and future life. Adults (parent, teacher, coach) expectations towards a child's abilities are consciously or unconsciously perceived by the child, influence his expectations of his own abilities, and thus his academic performance (Pygmalion effect). The child and his entourage's expectations are therefore a major factor to consider, especially in school-age children. According to ADHD studies, some brain areas involved in pain regulation and in attention cognitive abilities develop at a slower rate in children with ADHD than the other children.

Considering the deleterious consequences generated by the symptoms of this disorder, the research project aims to better understand the role of expectations in children with ADHD in a medical (pain) and school (attention abilities) context. It also aims to contribute to better understand the role of the brain on the expectations effect and ADHD. In this study, children expectations will be modulated while pain experiments and cognitive task will be realized by children with and without ADHD. Brain measures will also be assessed with advanced techniques.

Thus, we hope that the results will help improve intervention strategies in these contexts to ensure better support for children with ADHD, with a distant goal of contributing to the development of stronger tools for differential diagnostics.

DETAILED DESCRIPTION:
Attention Deficit with or without Hyperactivity Disorder (ADHD) is a neurodevelopmental disorder that affects 2 to 7% worldwide youth population and 6.2% of children aged 6 to 11 years in Quebec [1-3]. The main symptoms of this disorder are difficulties in regulating behaviour and/or concentration [4]. These difficulties have significant negative consequences in someone's life, particularly in terms of their academic success [5] and has significant negative consequences in the medical context, increasing accidents and mortality risk [6].

Children's academic performance can be modulated by the Pygmalion (or Rosenthal) effect, which refers to an improvement or decrease in an individual's performance depending on the degree of belief in his or her abilities on the part of an authority or the environment [7]. Thus, these beliefs have an influence on a person's expectations of his or her ability to do a task, and thus on final performance [8]. The expectations of an individual and his or her entourage is therefore a major factor to consider, especially in school-age children [9]. Expectations also play an important role in the placebo effect. Whereas a placebo is a treatment without any real influence on a particular condition (drug or therapeutic technique), the placebo effect is the perceived beneficial effect following this treatment. Furthermore, a placebo effect is almost always added to the beneficial effect of a treatment in different ways (for example, an analgesic effect could occur faster or in a shorter delay) and to different degrees [10]. The placebo effect is regularly studied and increasingly understood in the context of pain [11]. Although the perception of pain is influenced by placebo treatment, this effect is itself modulated by the expectations of the person in pain [12]. The dorsolateral prefrontal cortex (DLPFC) is an essential region for the placebo's mechanism of action [10]. In children with ADHD, there is a delay in the maturation of the cortical thickness of DLPFC between the ages of 7 and 10 years [13]. These differences in neuronal activity in the prefrontal region are associated with difficulties in attention control and inhibition in these children: inhibitory functions measured using transcranial magnetic stimulation (TMS) show a lower inhibition capacity in individuals with ADHD than without ADHD [14].

Considering the important consequences generated by the symptoms of this disorder, it is essential to better understand the role of the placebo/nocebo effect and expectations in children with ADHD in a medical (pain) and academic (attentional skills) context. Our goal is to better understand how this placebo/nocebo effects and expectations are associated with changes in the DLPFC and the inhibitory functions. This study also aims to better characterize the role of neurophysiological and neuroanatomical factors in these contexts, with the distant goal of contributing to the development of stronger tools for differential diagnostics.

Objectives (1) To compare the placebo/nocebo effect on pain and (2) on attention abilities in children with and without ADHD. (3) To determine if there is a relationship between the placebo/nocebo effect and neurophysiological (inhibitory mechanisms) and neuroanatomical (DLPFC) measures.

Assumptions

(1) Children with ADHD will have a weaker response to the placebo/nocebo effect on pain and (2) on attention abilities than children without ADHD (3) There is a moderate to strong association between the placebo/nocebo effect and neurophysiological/ neuroanatomical markers.

Methodology Data will be collected from 44 children, 22 with ADHD and 22 without ADHD.

At the first session, we will proceed with the experimentation of the placebo and nocebo effect on pain and on the ability to perform cognitive tasks. The experiment will be divided into two parts; a placebo part where the participant will have to take a "drug" (inactive; placebo) that improves cognitive abilities and pain tolerance for a short period of time, and a nocebo part where the participant will have to take a "drug" (inactive; nocebo) that decreases cognitive abilities and pain tolerance for a short period of time. The placebo/nocebo effect will be induced using an inactive capsule that "increases" or "reduces" (depending on the experimenter's discourse) general cognitive skills, as well as sensitivity and tolerance to pain. Following the administration of each capsule, we will proceed with the pain and attention experiments, all in a randomized order. Between the two parts of the experimentation, we will proceed to the questionnaire administration with the participant. Since all the steps are approximately 45 minutes in length, we will be able to plan a session with participants lasting between one and one and a half hours.

In the second session, we will perform the neurophysiological (inhibitory mechanisms) and neuroanatomical (DLPFC) measures. At the end of the visit, we will also proceed with a review of the study in order to disclose the information that was obscured during the project. An explanatory document containing this information and the participant's detailed participation will also be given to the parent and the child.

Analyses T-tests will be used to assess the effect of expectations on pain in children with ADHD compared to children without ADHD (Objective 1). The same analyses will be conducted to compare the effect of expectations on the ability to perform attentional cognitive tasks between the two groups (objective 2). For objective 3, simple regressions will first be used to determine whether there is an association between independent variables (neurophysiological and neuranatomical measures) and the effect of expectations on pain and cognitive tasks. Potentially predictive variables with a p-value ˂ 0.15 on the correlation test will be retained for the development of the multiple regression model. All possible models, and therefore all subsets of the variables retained in the previous step, will be considered. Statistical criteria (R2, adjusted R2 and Mallow's Cp) as well as a critical clinical judgment will allow us to decide on the best model. This final model will only include variables with a beta coefficient that is significantly non-zero at the alpha level of 0.05.

Non-parametric analyses will also be performed to determine if significant results can be obtained. In addition to providing preliminary results, this study will provide the statistical parameters (mean, standard deviation) required to calculate the sample size.

Contributions Research. This study could contribute to a better understanding of the role of expectations in children with ADHD, in a medical (pain) and academic (attentional skills) context. It will also allow us to better understand the role of DLPFC in the mechanism of the placebo/nocebo effect.

Clinic. As a result, it will be potentially possible to improve the intervention strategies to be implemented in order to ensure better support for children with ADHD, also in the medical (pain) and school (attentional skills) contexts. This study may also allow a better general understanding and evaluation of the disorder, and thus reduce prejudice towards children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Child 8 or 9 years old
* ADHD diagnosis confirmed by a qualified health professional (for the ADHD group only).
* Understand French

Exclusion Criteria:

* Other neurological problems other than ADHD
* Diagnosis of a psychological disorder
* Intellectual disability

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Placebo and nocebo effect on pain | Change from pre-test pain sensation to the pain sensation after the two "medications" (collected in one visit in March-April during the pre-test, after the placebo and after the nocebo. Data will be reported within the following 6 months.
  Pain (thermal) will be generated using an experimental pain paradigm using a thermode (heat). Perceived pain level will be assessed using a standardized tool; a computer-connected Visual Analogue Scale (VAS). The participant can score the pain sensation with a 0 to 10 scale, where 0 means "no pain" and 10 "the most intense pain tolerable".
Placebo and nocebo effect on attention abilities | Change from pre-test results to the results observed after the two "medications" (collected in one visit in March-April during the pre-test, after the placebo and after the nocebo. Data will be reported within the following 6 months.
  Attention abilities will be assessed using equivalent randomly assigned attentional tasks, the Stop signal task (SST). The measured outcomes are the reaction times in milisecond (ms) and the proportion of correct/incorrect reactions.

SECONDARY OUTCOMES:
Neuroanatomical measures : DLPFC gray matter volume | The outcome measure should be assessed during the visit 2, which should occur in 3-4 months. Data should be reported within the following 6 months.
  The neuroanatomy measurements will be assessed using magnetic resonance imaging (MRI). Structural MRI will be used to measure the DLPFC anatomy.
Neuroanatomical measures : DLPFC neural activity | The outcome measure should be assessed during the visit 2, which should occur in 3-4 months. Data should be reported within the following 6 months.
  The neuroanatomy measurements will be assessed using magnetic resonance imaging (MRI). Fonctionnal MRI will be used to measure the DLPFC neural activity.
Neuroanatomical measures : DLPFC neural connection | The outcome measure should be assessed during the visit 2, which should occur in 3-4 months. Data should be reported within the following 6 months.
  The neuroanatomy measurements will be assessed using magnetic resonance imaging (MRI).
  Diffusion MRI will be used to measure the DLPFC neural pathways.
Neuroanatomical measures : DLPFC vascularisation | The outcome measure should be assessed during the visit 2, which should occur in 3-4 months. Data should be reported within the following 6 months.
  The neuroanatomy measurements will be assessed using magnetic resonance imaging (MRI). Vascular MRI will be used to measure the DLPFC vascular network.
Neurophysiological measures: inhibitory mechanisms | The outcome measure should be assessed during the visit 2, which should occur in 3-4 months. Data should be reported within the following 6 months.
  The inhibitory mechanisms will be evaluated using transcranial magnetic stimulation (TMS) using the short intracortical interval inhibition measurement technique (short inhibition intracortical interval, SICI), were magnetic pulses are applied to the motor cortex. This method requires a double stimulation at an interval of 1 to 6 ms so that the muscle response usually observed is inhibited.
Heart rate measures | Change from pre-test results and to the results observed after the two "medications" (collected continuously in visit 1 in March-April during the pre-tests, after the placebo and after the nocebo. Data will be reported within the following 6 months.
  Heart rate measures will be collected with an electrocardiogram (using 3 electrodes in the back).
ADHD symptoms | Assessment during visit 1 in March-April. Data will be reported within the following 6 months.
  More information about the ADHD related symptoms and impacts will be collected by questionnaires for the parent.
Pain catastrophizing | Assessment during visit 1 in March-April. Data will be reported within the following 6 months.
  This data will be collected with the Pain Catastrophizing Scale for Children in French (PCS-C-FR). Scale from 0 to 52, where 0 is better and 52 is worse.
Anxiety traits | Assessment during visit 1 in March-April. Data will be reported within the following 6 months.
  This data will be collected with the State-Trait Anxiety Inventory for Children (STAI-CH)
Sleep quality - Child | Assessment during visit 1 in March-April. Data will be reported within the following 6 months.
  This data will be collected with the Morningness-Eveningness for Children Scale in French.
Sleep quality - Parent | Assessment during visit 1 in March-April. Data will be reported within the following 6 months.
  This data will be collected with the Pediatric Sleep Questionnaire in French (parent).
Sociodemographic measures | Assessment during visit 1 in March-April. Data will be reported within the following 6 months.
  This data will be collected with an adapted version of the the Canadian ADHD Ressource Alliance (CADDRA) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume guillaume.leonard2@usherbrooke.ca, pht., PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche sur le vieillissement (CdRV), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The final results will be shared in the published articles following the end of the study

REFERENCES:
- [Background] Polanczyk G, de Lima MS, Horta BL, Biederman J, Rohde LA. The worldwide prevalence of ADHD: a systematic review and metaregression analysis. Am J Psychiatry. 2007 Jun;164(6):942-8. doi: 10.1176/ajp.2007.164.6.942. PMID 17541055
- [Background] Sayal K, Prasad V, Daley D, Ford T, Coghill D. ADHD in children and young people: prevalence, care pathways, and service provision. Lancet Psychiatry. 2018 Feb;5(2):175-186. doi: 10.1016/S2215-0366(17)30167-0. Epub 2017 Oct 9. PMID 29033005
- [Background] Merten EC, Cwik JC, Margraf J, Schneider S. Overdiagnosis of mental disorders in children and adolescents (in developed countries). Child Adolesc Psychiatry Ment Health. 2017 Jan 17;11:5. doi: 10.1186/s13034-016-0140-5. eCollection 2017. PMID 28105068
- [Background] Janiaud P, Cornu C, Lajoinie A, Djemli A, Cucherat M, Kassai B. Is the perceived placebo effect comparable between adults and children? A meta-regression analysis. Pediatr Res. 2017 Jan;81(1-1):11-17. doi: 10.1038/pr.2016.181. Epub 2016 Sep 20. PMID 27648807
- [Background] Rainville P, Bao QVH, Chretien P. Pain-related emotions modulate experimental pain perception and autonomic responses. Pain. 2005 Dec 5;118(3):306-318. doi: 10.1016/j.pain.2005.08.022. Epub 2005 Nov 14. PMID 16289802
- [Background] Price DD, Finniss DG, Benedetti F. A comprehensive review of the placebo effect: recent advances and current thought. Annu Rev Psychol. 2008;59:565-90. doi: 10.1146/annurev.psych.59.113006.095941. PMID 17550344
- [Background] Benedetti F, Pollo A, Lopiano L, Lanotte M, Vighetti S, Rainero I. Conscious expectation and unconscious conditioning in analgesic, motor, and hormonal placebo/nocebo responses. J Neurosci. 2003 May 15;23(10):4315-23. doi: 10.1523/JNEUROSCI.23-10-04315.2003. PMID 12764120
- [Background] Friedman LA, Rapoport JL. Brain development in ADHD. Curr Opin Neurobiol. 2015 Feb;30:106-11. doi: 10.1016/j.conb.2014.11.007. Epub 2014 Dec 9. PMID 25500059
- [Background] Bruckmann S, Hauk D, Roessner V, Resch F, Freitag CM, Kammer T, Ziemann U, Rothenberger A, Weisbrod M, Bender S. Cortical inhibition in attention deficit hyperactivity disorder: new insights from the electroencephalographic response to transcranial magnetic stimulation. Brain. 2012 Jul;135(Pt 7):2215-30. doi: 10.1093/brain/aws071. Epub 2012 Apr 3. PMID 22492560
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] McGrath PA, Seifert CE, Speechley KN, Booth JC, Stitt L, Gibson MC. A new analogue scale for assessing children's pain: an initial validation study. Pain. 1996 Mar;64(3):435-443. doi: 10.1016/0304-3959(95)00171-9. PMID 8783307
- [Background] Kujirai T, Caramia MD, Rothwell JC, Day BL, Thompson PD, Ferbert A, Wroe S, Asselman P, Marsden CD. Corticocortical inhibition in human motor cortex. J Physiol. 1993 Nov;471:501-19. doi: 10.1113/jphysiol.1993.sp019912. PMID 8120818